CLINICAL TRIAL: NCT06711679
Title: Exploring the Minimum Effective Concentration and Volume of Ropivacaine for Sacral Plexus Anesthesia in Children of Different Ages
Brief Title: Exploring the Minimum Effective Concentration and Volume of Ropivacaine for Sacral Plexus Anesthesia
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Yilin Zhao (Other)
Collaborators: Henan Provincial People's Hospital (Other); Wuhan Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yilin Zhao, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024S006
Record Dates: First submitted 2024-11-19; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Pediatric ALL
Keywords: Caudal anesthesia; Children; Thermal imaging; Intraoperative MRI
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Ropivacaine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neonatal group (Experimental): From birth to 28 days
  Interventions: Drug: Low-dose ropivacaine; Drug: Medium-dose of ropivacaine; Drug: High-dose ropivacaine
- Infant group (Experimental): 1 month to 1 year
  Interventions: Drug: Low-dose ropivacaine; Drug: Medium-dose of ropivacaine; Drug: High-dose ropivacaine
- Toddler Group (Experimental): 1-3 years
  Interventions: Drug: Low-dose ropivacaine; Drug: Medium-dose of ropivacaine; Drug: High-dose ropivacaine
- Child Group (Experimental): 3-7 years
  Interventions: Drug: Low-dose ropivacaine; Drug: Medium-dose of ropivacaine; Drug: High-dose ropivacaine

INTERVENTIONS:
Drug: Low-dose ropivacaine — 0.5 ml/Kg ropivacaine
  Other Names: MRI scan
Drug: Medium-dose of ropivacaine — 1ml/Kg ropivacaine
  Other Names: MRI scan
Drug: High-dose ropivacaine — 1.5 ml/Kg ropivacaine
  Other Names: MRI scan

SUMMARY:
The goal of this clinical trial is to explore the minimum effective concentration and volume of ropivacaine for sacral plexus anesthesia. The main questions it aims to answer are:

* The distribution of different volumes of ropivacaine after caudal anesthesia
* The blockade level after caudal anesthesia with varying doses
* The minimum effective concentration of ropivacaine among pediatric patients of different age groups Researchers will inject different doses or concentrations of ropivacaine into the caudal canal to observe the drug's spread range, the level of blockade, and the duration of its effect.

Participants will:

* Undergo magnetic resonance imaging (MRI) examinations before and after caudal anesthesia
* Will be detected the blockade level after caudal anesthesia

DETAILED DESCRIPTION:
The activity of CYP1A2 in newborns and infants is lower than in adults, which may result in slower metabolism of ropivacaine. This might necessitate a reduction in the dosage or concentration of ropivacaine to prevent drug accumulation and toxicity. Additionally, since the nervous system in children is still developing, excessively high concentrations of ropivacaine could have adverse effects. Therefore, the lowest effective concentration of ropivacaine should be chosen to minimize the risk of adverse reactions. Generally, the dosage of ropivacaine should be determined based on the patient's age, weight, and the type of surgery. However, there are currently no definitive dosage recommendations, and further research is needed to determine these guidelines.

The goal of this clinical trial is to exploring the minimum effective concentration and volume of ropivacaine for sacral plexus anesthesia. Using MRI to investigate the distribution of different doses of ropivacaine after caudal anesthesia, and employing infrared imaging technology to detect the blockade level after caudal anesthesia with varying doses.

Participants will receive 0.5ml/Kg, 1ml/Kg and 1.5ml/Kg ropivacaine, then undergo magnetic resonance imaging (MRI) examinations to detect the distribution and optic nerve sheath diameter (ONSD) before and after caudal injection. Also, the blockade level will be detected 15min and 30 min after caudal anesthesia

ELIGIBILITY:
Inclusion Criteria:

BMI ≤ 30 kg/m²; lower limbs surgery; lower abdomen surgery; perineal region surgery; Normal liver and kidney function; Normal coagulation function; Hemoglobin > 70 g/L.

Exclusion Criteria:

Abnormal coagulation function; Allergy to local anesthetics; Abnormal sacral anatomy; Puncture site infection;

Ages: 1 Day to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Distribution and block plane in the spinal canal after caudal injection of different doses of ropivacaine. | 30 minutes
  MRI scan will be performed before and after 0.5 ml/Kg, 1,ml/Kg, or 1.5ml/Kg ropivacaine injection,
The blockade level after caudal anesthesia with varying doses | 60 minutes
  The blockade level will be tested 15 min and 30min after 0.5 ml/Kg, 1,ml/Kg, or 1.5ml/Kg ropivacaine injection. The infrared imaging technology will be employed to test the blockade level.
The minimum effective concentration of ropivacaine among pediatric patients of different age groups | 2 days
  The fixed capacity requires the minimum effective concentration by changing the concentration

SECONDARY OUTCOMES:
Effects ofMedium-dose and high-dose of ropivacaine injection on Optic Nerve Sheath Diameter (ONSD) and blood brain barrier | 60 minutes
  Optic Nerve Sheath Diameter (ONSD) and blood brain barrier will be meseared before and after injection, and after sugery operation
Effects of different volumes and concentrations of ropivacaine on heart rate | 2 days
  Effects on heart rate after different volumes and concentrations of ropivacaine injection
Effects of different volumes and concentrations of ropivacaine on blood pressure | 2 days
  Effects on blood pressure after different volumes and concentrations of ropivacaine injection
Effects of different volumes and concentrations of ropivacaine on oxygenation | 2 days
  Effects on oxygenation after different volumes and concentrations of ropivacaine injection
To evaluate the relaxation degree of anal sphincter after sacral anesthesia | 30 minutes
  Measure the pressure changes of the anal sphincter after caudal anesthesia using a pressure sensor

CONTACTS AND LOCATIONS:
Overall Officials: Yilin Zhao, M.D, Ph.D, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No